CLINICAL TRIAL: NCT01565070
Title: Osteoarthritis in Older Adults: Recovery of Mobility and Pain With a Topical Analgesic
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The local authorities did not authorize the use of biofreeze in Chile.
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Daniel Bunout, Medical Doctor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIOFREEZE OSTEOARTHRITIS; HYGIENIC CORPORATION (Other Grant/Funding Number: HYGIENIC CORPORATION)
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2012-03

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Pain; Quality of life
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biofreeze (Active Comparator)
  Interventions: Drug: Biofreeze
- Placebo (Placebo Comparator): Use of placebo ointment
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Biofreeze — Use of Biofreeze ointment
  Arms: Biofreeze
Other: Placebo — Use of placebo ointment
  Arms: Placebo

SUMMARY:
Biofreeze® is a topical ointment that has menthol and alcamphor. Its analgesic effect lies in the stimulation of A and C fibers by cold and nociceptive stimulation, respectively, which is produced by menthol, apparently through the newly discovered receptor TRPM8 (Transient Receptor Potential melastatin-8) The aim of this study is to investigate if BIOFREEZE ® treatment (Performance Health Inc., Export, PA) improves symptoms associated with moderate knee osteoarthritis, which would decrease the immobility and isolation in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Moderate osteoarthritis of the knee
* Age 60 to 80 years
* Ambulatory

Exclusion Criteria:

* Other conditions that affect mobility
* Severe chronic diseases such as cardiac or renal failure
* Cancer
* Presence of gout
* Cognitive impairment

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
WOMAC score | 60 days
  WOMAC score corresponds to Western Ontario and McMaster Universities Index of Osteoarthritis

SECONDARY OUTCOMES:
Quality of life measured using SF 36 | 60 days
  SF 36 correponds to a health related quality of life score

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bunout, MD, Principal Investigator — INTA University of Chile
Locations (1):
- Institute of Nutrition and Food Technology, Santiago, Met, Chile

REFERENCES:
- [Background] Zhang J, Enix D, Snyder B, Giggey K, Tepe R. Effects of Biofreeze and chiropractic adjustments on acute low back pain: a pilot study. J Chiropr Med. 2008 Jun;7(2):59-65. doi: 10.1016/j.jcme.2008.02.004. PMID 19674721